CLINICAL TRIAL: NCT06059937
Title: Evaluation of Cardiovascular Risk After Preeclampsia in General Practitioners and Patients
Acronym: PreCarVasc
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Marc BOIVIN, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2023-A00933-42
Record Dates: First submitted 2023-06-20; First posted 2023-09-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Patients Hospitalized for Pre-eclampsia
Keywords: pre-eclampsia; cardiovascular risk
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Patient with pre-eclampsia — Cardiovascular risk assessment by the general practitioner in the year following pre-eclampsia

SUMMARY:
Pre-eclampsia is a disease characterized by placental damage leading to a cascade of complications during pregnancy. It is initially manifested by high blood pressure and the presence of albumin in the urine. It can lead to emergency hospitalization in severe cases and cause major complications or even death in the mother and the fetus.

Several studies observing the outcome of patients with pre-eclampsia have shown an increased long-term cardiovascular risk in these patients, justifying regular medical follow-up with the treating physician and specialists, mainly cardiologists.

The main objective of this research is to describe the cardiovascular risk assessment actions implemented by the treating general practitioner in the year following pre-eclampsia (blood pressure measurement in the office, self-measurement of blood pressure, ABPM, cardiological consultation, biological monitoring of blood (creatininemia, LDL, fasting glycemia) or urine (albuminurie/creatininurie ratio), and screening and management of possible smoking).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years hospitalized for preeclampsia at the Nancy regional maternity hospital

Exclusion Criteria:

* Fetal death in utero;
* Adult Person subject to a legal protection measure (guardianship, curatorship, safeguard of justice);
* Person deprived of liberty by a judicial or administrative decision;
* Person subject to psychiatric care under constraint by virtue of articles L. 3212-1 and L. 3213-1 of the Public Health Code.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years of age who were hospitalized for preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Performing a blood pressure measurement by the general practitioner | Up to one year following pre eclampsia
  Description: Describe the cardiovascular risk assessment actions implemented by the general practitioner in the year following pre-eclampsia within the following specific monitoring tools such as blood pressure measurement in the office. Composite outcome with 2, 3, 4, 5 and 6
Performing a self-measurement of blood pressure | Up to one year following pre eclampsia
  Description: Describe the cardiovascular risk assessment actions implemented by the general practitioner in the year following pre-eclampsia within the following specific monitoring tools such as self-measurement of blood pressure. Composite outcome with 2, 3, 4, 5 and 6
Performing a cardiological consultation | Up to one year following pre eclampsia
  Description: Describe the cardiovascular risk assessment actions implemented by the general practitioner in the year following pre-eclampsia within the following specific monitoring tools such as cardiological consultation. Composite outcome with 2, 3, 4, 5 and 6
Performing a ambulatory measurement of blood pressure | Up to one year following pre eclampsia
  Description: Describe the cardiovascular risk assessment actions implemented by the general practitioner in the year following pre-eclampsia within the following specific monitoring tools such as ambulatory measurement of blood pressure. Composite outcome with 2, 3, 4, 5 and 6
Performing a biological monitoring of blood (creatinine, LDL cholesterol, fasting glucose, albuminuria creatinuria ratio) | Up to one year following pre eclampsia
  Description: Describe the cardiovascular risk assessment actions implemented by the general practitioner in the year following pre-eclampsia within the following specific monitoring tools such as biological monitoring of blood (creatinine, LDL, fasting glucose) or urine (Albuminuria/creatininuria ratio). Composite outcome with 2, 3, 4, 5 and 6.
Screening and management of possible smoking | Up to one year following pre eclampsia
  Description: Describe the cardiovascular risk assessment actions implemented by the general practitioner in the year following pre-eclampsia within the following specific monitoring tools such as screening and management of possible smoking. Composite outcome with 1, 2, 3, 4 and 5

SECONDARY OUTCOMES:
Cardiovascular risk assessment by the general practitioner | Up to 5 years following pre eclampsia
  Patient's cardiovascular risk evaluation by the general practitioner (low, medium, high or very high).
Cardiovascular risk assessment by the patient | Up to 5 years following pre eclampsia
  Patient's cardiovascular risk evaluation by the patient (low, medium, high or very high).
Knowledge of pre-eclampsia status | Up to 5 years following pre eclampsia
  Knowledge of the pre-eclampsia status of the patient by the general practitioner.
Pre eclampsia information mode | Up to 5 years following pre eclampsia
  How general practitioner is informed about pre-eclampsia
Performing a blood pressure measurement | Up to one year following pre eclampsia
  Actions implemented by the general practiotioner within the following specific tools as reported by the patient such as blood pressure measurement in the office.
Performing a self-measurement of blood pressure | Up to one year following pre eclampsia
  Actions implemented by the general practiotioner within the following specific tools as reported by the patient.such as self-measurement of blood pressure.
Performing a cardiological consultation | Up to one year following pre eclampsia
  Actions implemented by the general practiotioner within the following specific tools as reported by the patient such as cardiological consultation.
Performing a ambulatory measurement of blood pressure | Up to one year following pre eclampsia
  Actions implemented by the general practiotioner within the following specific tools as reported by the patient such as ambulatory measurement of blood pressure.
Performing a biological monitoring of blood (creatinine, LDL cholesterol, fasting glucose, albuminuria creatinuria ratio) | Up to one year following pre eclampsia
  Actions implemented by the general practiotioner within the following specific tools as reported by the patient such as biological monitoring of blood (creatinine, LDL, fasting glucose) or urine (Albuminuria/creatininuria ratio).
Screening and management of possible smoking | Up to one year following pre eclampsia
  Actions implemented by the general practiotioner within the following specific tools as reported by the patient such as screening and management of possible smoking.
Rate of hypertension following pre-eclampsia | Up to 5 years following pre eclampsia
  Composite endpoint of hypertension, stroke and/or coronary accident with 17;18
Rate of stroke following pre-eclampsia | Up to 5 years following pre eclampsia
  Composite endpoint of hypertension, stroke and/or coronary accident with 16;18
Rate of coronary accident following pre-eclampsia | Up to 5 years following pre eclampsia
  Composite endpoint of hypertension, stroke and/or coronary accident with 16;17

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, MD-PhD, Study Chair — CHRU de NANCY
Locations (1):
- CHRU de NANCY, Vandœuvre-lès-Nancy, France